CLINICAL TRIAL: NCT01936610
Title: the Effect of Instructional Method on Decision Making
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zahra Abedian, Instructor of Midwifery, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: educational
Record Dates: First submitted 2013-09-03; First posted 2013-09-06 (Estimated); Last update posted 2013-09-06 (Estimated); Status verified 2010-05

CONDITIONS: Pregnancy
Keywords: Lecture; Role-playing; Knowledge; Attitude; Decision making; Type of delivery
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- role play (Experimental): In this method, researcher with two other co-researchers played 3 scenarios in 7 steps (for each scenario)including warm up, selecting participant, preparing the scene, preparing observers, play ,discussion and evaluation and generalization to education about advantages and disadvantages of normal delivery and cesarean section .
  Interventions: Other: role play
- lecture (Experimental): describe the advantages and disadvantages of normal delivery and cesarian section
  Interventions: Other: lecture

INTERVENTIONS:
Other: role play — In this method, researcher with two other co-researchers played 3 scenarios in 7 steps (for each scenario)including warm up, selecting participant, preparing the scene, preparing observers, play ,discussion and evaluation and generalization to education about advantages and disadvantages of normal delivery and cesarean section.
  Arms: role play
Other: lecture — Describe advantages and disadvantages in one 90-min session
  Arms: lecture

SUMMARY:
In these single- blind clinical trial 67 primigravida females, gestational aged 34-36 week were selected using multi-stage sampling and assigned into two groups randomly. Decision-making (before, two weeks after and at admission in maternity department) was tested by a researcher -made questionnaire. In experiment group, advantages and disadvantages of normal delivery and cesarean-section delivery were presented by role-playing in three 90-min scenarios. It was also presented in a 90-min lecture. Data were analyzed using SPSS by mean difference test, exact fisher test, independent t-test and paired t-test.

ELIGIBILITY:
Inclusion Criteria:

primipara , single pregnancy , gestational age of 34-36 weeks ,age of 18-35 years old, no history of infertility, no indication for cesarean section, no passing educational course for delivery methods

Exclusion Criteria:

medical condition in pregnant woman, diagnosis of abnormal fetus / no possibility for delivery fetus by sonography, abnormal volume of amniotic fluid or placenta

Ages: 20 Years to 28 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2010-06; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Decision making | 2 weeks
  Two weeks after educational course for each group (Lecture and Role play), knowledge, attitude and decision making questionnaire were completed again. They were followed at admission by phone conversation for knowing their decision.